CLINICAL TRIAL: NCT00078728
Title: Family-Based Prevention for Childhood Anxiety
Brief Title: Family-Based Prevention Program for Childhood Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K23MH063427 (NIH); K23MH063427 (NIH)
Record Dates: First submitted 2004-03-05; First posted 2004-03-08 (Estimated); Results first posted 2013-12-16 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-01

CONDITIONS: Anxiety Disorders
Keywords: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Family-based anxiety prevention program (Experimental): Participants will complete an 8 session (1 session/week), cognitive behavioral therapy-based, family prevention program to be administered by a trained clinician, after randomization to the study. The prevention program will include 3 booster sessions that take place after the first 8 sessions.
  Interventions: Behavioral: Family-Based Anxiety Prevention Program
- Evaluation only (Active Comparator): Waitlist control group. Participants in this group will receive general information (in the form of a printed packet) about anxiety after randomization to the study. Families in this group will complete all study evaluations and will then be offered the option of participating in the prevention program. Families who accept will begin the prevention sessions and will receive the same CBT-based, family-based prevention program as the other treatment arm.
  Interventions: Behavioral: Evaluation only

INTERVENTIONS:
Behavioral: Family-Based Anxiety Prevention Program — Participants in the prevention program will have weekly sessions with a therapist and will learn skills to help reduce anxiety for 8 weeks. The intervention will begin immediately after randomization to the study.
  Arms: Family-based anxiety prevention program
Behavioral: Evaluation only — Participants will undergo evaluations without active treatment for 8 weeks.
  Arms: Evaluation only

SUMMARY:
This study will evaluate the effectiveness of a short-term family-based program for preventing anxiety disorders in at-risk children.

DETAILED DESCRIPTION:
Anxiety disorders are serious conditions that can negatively impact a person's overall functioning. This study will enroll mothers with anxiety disorders and their children to determine whether a brief family-based intervention will reduce childhood anxiety better than standard care.

Participants will be randomly assigned to either the family-based prevention program or to evaluation only for 8 weeks. Participants in the prevention program will have weekly sessions with a therapist and will learn skills to help reduce anxiety. Self- and parent-reports, diagnostic interviews, a computerized memory task, and a videotaped parent-child interaction task will be used to assess participants. Assessments will be conducted at study start and one week after intervention completion (Week 9). Follow-up visits will be conducted at 6 and 12 months after intervention completion.

ELIGIBILITY:
Inclusion Criteria:

* Mothers with a current, primary anxiety disorder
* 7-12 year old children without an anxiety disorder

Exclusion Criteria:

* Mothers that do not have a current, primary anxiety disorder
* 7-12 year old children with an anxiety disorder
* 7-12 year old children that are currently receiving treatment for anxiety that could interfere with the study

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2003-09; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Golda S. Ginsburg, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 Family-based Prevention Program: Family-Based Anxiety Prevention Program : Participants in the prevention program will have weekly sessions with a therapist and will learn skills to help reduce anxiety for 8 weeks.
- 2 Evaluation Only: Evaluation only : Participants will undergo evaluations without active treatment for 8 weeks.
Period: Overall Study
Arm/Group | 1 Family-based Prevention Program | 2 Evaluation Only
Started | 20 | 20
Completed | 16 | 17
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Family-based Prevention Program | 2 Evaluation Only | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 20 | 40
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.20 (1.91) | 8.68 (1.81) | 8.94 (1.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 10 | 12 | 22
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Children With Child Anxiety Diagnosis
Description: Measured by the Anxiety Disorder Interview Schedule for the Diagnostic and Statistical Manual of Mental Disorders 4th edition, child and parent versions.
Time Frame: 12 month
Measure: Number; unit: participants
Groups:
- 2 Evaluation Only: Evaluation only : Participants will undergo evaluations without active intervention for 8 weeks but received an informational packet on anxiety disorders.
Arm/Group | 1 Family-based Prevention Program | 2 Evaluation Only
Number analyzed (Participants) | 20 | 20
participants | 20 | 20

2. Primary Outcome: Child Anxiety Diagnoses
Description: The cumulative number of children who developed an anxiety disorder at each assessment point during the study. Using the intent to treat sample, a total of 6 children in the non-intervention group developed an anxiety disorder by the 12-month assessment. No children in the CAPS group developed an anxiety disorder.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | 1 Family-based Prevention Program | 2 Evaluation Only
Number analyzed (Participants) | 20 | 20
participants | 0 | 6

ADVERSE EVENTS:
Arm/Group | 1 Family-based Prevention Program | 2 Evaluation Only
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
Of the 40 participants in the study, no adverse events occured or were reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No